CLINICAL TRIAL: NCT02773901
Title: Comparison of the Non-invasive ICP HeadSense Monitor vs Lumbar CSF Pressure Measurement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HeadSense Medical (Industry)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-031
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2016-12

CONDITIONS: Intracranial Hypertension
Keywords: intracranial pressure; noninvasive monitoring; lumbar puncture
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): ICP monitoring will be done with the HS-1000 to compare to CSF measurement from lumbar puncture (per clinical protocol without any change in the patient's management). HS-1000 ICP monitoring intervals last 10 minutes.
  Interventions: Device: HS-1000

INTERVENTIONS:
Device: HS-1000

SUMMARY:
In current practice patients with a suspected increase of intracranial pressure (ICP) will undergo a lumbar puncture with measurement of cerebral spinal fluid (CSF) pressure (as a marker for ICP). A lumbar puncture is an invasive and sometimes painful procedure. Using a new type of ICP monitor (HeadSense) it is possible to measure ICP non-invasively through an acoustic signal

DETAILED DESCRIPTION:
In this study we will prospectively collect relevant clinical data on 60 neurological patients, who are being referred for an elective lumbar puncture (eg. suspected multiple sclerosis, raised intracranial hypertension, etc). Each enrolled patient will be monitored in parallel to the lumbar puncture with the HeadSense ICP monitor. Subjects who meet the study inclusion and exclusion criteria will be enrolled in the study.

Step 1: 10 minute measurement of HeadSense monitor. Once the patient is inclined with his upper body 30 degrees to the bed the pressure values, the clinical procedure can begin. The device must be preset in a continuous monitoring mode. The continuous monitoring allows a loop of measurements for an unlimited time in a rate of four measurements per minute.

Step 2: 10 minute measurement of HeadSense monitor in supine position.

Step 3: Patient will be placed in a left lateral position. The lumbar puncture will be done and CSF pressure will be measured following standard procedures.

Step 4: 10 minute measurement of HeadSense monitor in supine position.

Lumbar puncture and HeadSense measurement will be done by two different doctors and they will not share measurement values during the procedure.

After the study the patient's ears will be examined for internal ear infection or irritation that might be caused by the ear buds. Patient adverse events will be documented on the case report forms in case they occurred and the family or advocate of the patient will be informed. In case of clinical relevant adverse events appropriate clinical action will be taken.

As the procedure does not affect the patient management, there is no need to provide any specific medical care related to the trial. Patients will receive the relevant clinical care related to their clinical management, without any consideration to their participation in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female in the age range of 18 years and older
* All patients who are referred for elective or subacute lumbar puncture including CSF pressure measurement

Exclusion Criteria:

* Local infection in the ear
* Pregnant or lactating women
* Cervical spine stenose
* Arnold-Chiari malformations
* Aqueductal stenosis or other changes causing an uneven CSF pressure between different compartments
* Mass lesions
* Current or previous craniotomy or craniectomies
* Suspicion of meningitis or encephalitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of ICP values obtained by the HeadSense device that correlate to ICP using current standards | 10 minutes

SECONDARY OUTCOMES:
Incidence of Adverse events (AEs) | 48 hours from the end of monitoring with the HS-1000

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schytz, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (3):
- Rigshospitalet-Glostrup, Copenhagen, Denmark
- Asklepios Hospitals Schildautal, Seesen, Germany
- Elisabeth/Tweesteden Hospital, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: No